CLINICAL TRIAL: NCT01034397
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess Efficacy of Tocilizumab+Non-biological DMARD in Reducing Synovitis as Measured by MRI at 12 Weeks After Initiation of Treatment in Patients With Moderate to Severe Rheumatoid Arthritis With Inadequate Response to Non-biological DMARDs
Brief Title: A Study of Tocilizumab Plus Non-biological DMARD in Patients With Moderate to Severe Rheumatoid Arthritis and an Inadequate Response to Non-biological DMARDs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML22648; 2009-012218-30
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: non-biological DMARDs
- 2 (Placebo Comparator)
  Interventions: Drug: placebo; Drug: non-biological DMARDs

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg (minimal dose 480mg, maximum dose 800mg) iv infusion every 4 weeks for 24 weeks
  Arms: 1
Drug: placebo — iv every 4 weeks for 24 weeks
  Arms: 2
Drug: non-biological DMARDs — stable dose at investigator's prescription

SUMMARY:
This randomized, double-blind, placebo-controlled study will use Magnetic Resonance Imaging (MRI) to assess the efficacy of tocilizumab plus non-biological DMARD in patients with moderate to severe rheumatoid arthritis who have had an inadequate response to non-biological DMARDS. Patients will be randomized to receive either intravenous tocilizumab at 8mg/kg (minimal dose 480mg, maximum dose 800mg) or placebo every 4 weeks, in addition to their stable dose of non-biological DMARD. Anticipated time on study treatment is 24 weeks, and target sample size is <100.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* moderate to severe rheumatoid arthritis of >/=6 months duration
* synovitis (swollen and tender joint) in the wrist of the dominant hand
* non-biologic DMARDs at stable dose for >/=12 weeks prior to baseline
* oral corticosteroids at stable dose for at least 25 out of 28 days prior to baseline

Exclusion Criteria:

* rheumatic autoimmune disease other than RA
* history of or current inflammatory joint disease other than RA
* functional class IV (ACR classification)
* intraarticular or parenteral corticosteroids within 6 weeks prior to baseline
* previous treatment with a biologic agent for RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Portugal (6):
  - Almada
  - Coimbra
  - Lisbon
  - Ponte de Lima
  - Porto
  - Vila Nova de Gaia

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 Milligrams Per Kilogram (mg/kg): Participants received tocilizumab 8 mg/kg (minimum dose of 480 mg, maximum dose of 800 mg) intravenously (IV) once every 4 weeks for 24 weeks.
- Placebo: Participants received placebo IV once every 4 weeks for a maximum of 24 weeks. At 12 weeks, participants who did not respond to treatment (those who did not show improvement of greater than or equal to [≥]20 percent [%] in tender joint count and swollen joint count) were offered rescue therapy with open-label tocilizumab 8 mg/kg every 4 weeks through Week 24.
Period: Overall Study
Arm/Group | Tocilizumab 8 Milligrams Per Kilogram (mg/kg) | Placebo
Started | 35 | 19
Completed | 28 | 17
Not Completed | 7 | 2
Not completed — Lack of compliance | 0 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to Treat (ITT) population: all participants randomized who had at least one efficacy measurement performed.
Groups:
- Placebo: Participants received placebo IV once every 4 weeks for a maximum of 24 weeks. At 12 weeks, participants who did not respond to treatment (those who did not show improvement of ≥20% in tender joint count and swollen joint count) were offered rescue therapy with open-label tocilizumab 8 mg/kg every 4 weeks through Week 24.
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg (minimum dose of 480 mg, maximum dose of 800 mg) IV once every 4 weeks for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tocilizumab 8 mg/kg | Total
Number analyzed (Participants) | 19 | 35 | 54
Age, Continuous [Median (Full Range); unit: years] | 54 [45 to 69] | 54 [28 to 79] | 54 [28 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 29 | 46
  Male | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Synovitis Measured by Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Score
Description: Synovitis is defined as an area in the synovial compartment that shows above normal postgadolinium enhancement of a thickness greater than the width of the normal synovium. T1-weighted images were acquired before and after the administration of intravenous contrast agent containing gadolinium. Intravenous contrast was required to demonstrate enhancing synovitis. Three wrist regions (distal radioulnar joint, radiocarpal joint, the intercarpal and intermetacarpal joint) and the 2nd to 5th metacarpophalangeal (MCP) were assessed for synovitis via magnetic resonance imaging (MRI) and scored using a scale ranging from 0-3 where 0 is normal and scores 1-3 (mild, moderate, severe) are by thirds of the presumed volume of enhancing tissue in the synovial compartment. These values were then summed yielding scores of 0-9 in the wrist region, 0-12 for MCP joints, and 0-22 on the aggregate. A negative value in synovitis change from Baseline score indicates an improvement.
Time Frame: Week 12
Population: ITT population; n (number) equals (=) number of participants assessed for the specified parameter
Measure: Median (Full Range); unit: percent change
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg (minimum dose of 480 mg, maximum dose of 800 mg) IV once every 4 weeks for 20 weeks (total of 6 infusions).
- Placebo: Participants received placebo IV once every 4 weeks for a maximum of 20 weeks (total of 6 infusions). At 12 weeks, participants who did not respond to treatment (those who did not show improvement of ≥20% in tender joint count [TJC] and swollen joint count [SJC]) were offered rescue therapy with open-label tocilizumab 8 mg/kg IV once every 4 weeks through Week 20.
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
percent change
  Wrist region (n=30,17) | -20.0 [-100.0 to 200.0] | -37.5 [-100.0 to 40.0]
  2nd to 5th MCP joints (n=25,14) | -25.0 [-91.7 to 100.0] | 0.0 [-100.0 to 100.0]
  Total synovitis score (n=30,17) | -23.6 [-80.0 to 1200.0] | -25.0 [-69.2 to 60.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided — Wrist region: Tocilizumab versus placebo; Since one-sided t-test was used all effects in the opposite direction of what was predicted have a p-value=1
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.026, t-test, 1 sided — 2nd and 5th MCP joints: Tocilizumab versus placebo
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided — Total synovitis score: Tocilizumab versus placebo; Since one-sided t-test was used all effects in the opposite direction of what was predicted have a p-value=1

2. Secondary Outcome: Percent Change From Baseline to Week 12 in OMERACT RAMRIS Score
Description: RAMRIS score is the sum of its core components: Synovitis Score, Edema Score, and Erosion Score. Synovitis scored from 0 (normal) to 9 (maximum distension of synovial cavity). Edema scored 0 (normal) to 69 (maximum articular bone involvement). Erosion scored from 0 (normal) to 230 (maximum erosion of articular bone). RAMRIS=Synovial Score plus (+) Edema Score + Erosion Score. Minimum RAMRIS score=0 (normal), maximum RAMRIS score=308 (severe structural damage). For Synovial Score, Edema Score, Erosion Score, and RAMRIS score, increasing number=increasing severity.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: percent change
Groups:
- Placebo: Participants received placebo IV once every 4 weeks for a maximum of 20 weeks (total of 6 infusions). At 12 weeks, participants who did not respond to treatment (those who did not show improvement of ≥20% in TJC and SJC) were offered rescue therapy with open-label tocilizumab 8 mg/kg IV once every 4 weeks through Week 20.
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
percent change | -10.6 [-80.9 to 127.8] | -15.4 [-59.7 to 41.7]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.421, t-test, 1 sided — Percentage Change in OMERACT RAMRIS global score; Tocilizumab versus placebo

3. Secondary Outcome: Absolute Change From Baseline to Week 12 in OMERACT RAMRIS Score
Description: as for outcome 2
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
units on a scale | -5.5 [-38.0 to 23.0] | -7.0 [-43.0 to 15.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.434, t-test, 1 sided — Absolute change in OMERACT RAMRIS global score; Placebo versus Tocilizumab

4. Secondary Outcome: Percent Change From Baseline to Week 24 in OMERACT RAMRIS Score
Description: RAMRIS score is the sum of its core components: Synovitis Score, Edema Score, and Erosion Score. Synovitis scored from 0 (normal) to 9 (maximum distension of synovial cavity). Edema scored 0 (normal) to 69 (maximum articular bone involvement). Erosion scored from 0 (normal) to 230 (maximum erosion of articular bone). RAMRIS=Synovial Score + Edema Score + Erosion Score. Minimum RAMRIS score=0 (normal), maximum RAMRIS score=308 (severe structural damage). For Synovial Score, Edema Score, Erosion Score, and RAMRIS score, increasing number=increasing severity.
Time Frame: Week 24
Population: ITT population; participants from the placebo group who did not show an improvement of ≥20% in TJC and SJC were offered recovery therapy with tocilizumab 8 mg/kg and were placed in Placebo-Tocilizumab 8 mg/kg group.
Measure: Median (Full Range); unit: percent change
Groups:
- Placebo: Participants received placebo IV once every 4 weeks for a maximum of 20 weeks (total of 6 infusions).
- Placebo-Tocilizumab 8 mg/kg: Participants received placebo IV once every 4 weeks for 12 weeks (total of 3 infusions). At 12 weeks, participants who did not respond to treatment (those who did not show improvement of ≥20% in TJC and SJC) received tocilizumab 8 mg/kg IV once every 4 weeks through Week 20.
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 7 | 9
percent change | -24.2 [-70.0 to 83.3] | -17.3 [-33.3 to -4.2] | -36.8 [-73.7 to 11.8]

5. Secondary Outcome: Absolute Change From Baseline to Week 24 in OMERACT RAMRIS Score
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 4
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 7 | 9
units on a scale | -13.0 [-34.0 to 15.0] | -3.0 [-24.0 to -1.0] | -14.0 [-46.0 to 4.0]

6. Secondary Outcome: Absolute Change From Baseline to Week 12 in OMERACT-RAMRIS Synovitis Score
Description: Synovitis is defined as an area in the synovial compartment that shows above normal postgadolinium enhancement of a thickness greater than the width of the normal synovium. T1-weighted images were acquired before and after the administration of intravenous contrast agent containing gadolinium. Intravenous contrast was required to demonstrate enhancing synovitis. Three wrist regions (distal radioulnar joint, radiocarpal joint, the intercarpal and intermetacarpal joint) and the 2nd to 5th MCP were assessed for synovitis via MRI and scored using a scale ranging from 0-3 where 0 is normal and scores 1-3 (mild, moderate, severe) are by thirds of the presumed volume of enhancing tissue in the synovial compartment. These values were then summed yielding scores of 0-9 in the wrist region, 0-12 for MCP joints, and 0-22 on the aggregate. A negative value in synovitis change from Baseline score indicates an improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
units on a scale
  Wrist region | -1.0 [-6.0 to 3.0] | -2.0 [-8.0 to 2.0]
  2nd to 5th MCP joints | -1.0 [-11.0 to 10.0] | 0.0 [-4.0 to 6.0]
  Total synovitis score | -2.0 [-14.0 to 12.0] | -2.0 [-9.0 to 5.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided — Change in Wrist region; Tocilizumab versus placebo. Since one-sided t-test was used all effects in the opposite direction of what was predicted have a p-value=1
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.065, t-test, 1 sided — Change in 2nd to 5th MCP; Tocilizumab versus placebo
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided — Change in Total synovitis; Tocilizumab versus placebo. Since one-sided t-test was used all effects in the opposite direction of what was predicted have a p-value=1

7. Secondary Outcome: Absolute Change From Baseline to Week 24 in OMERACT-RAMRIS Synovitis Score
Description: as for outcome 6
Time Frame: Week 24
Population: ITT population.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 7 | 9
units on a scale
  Wrist region | -1.0 [-7.0 to 2.0] | -2.0 [-5.0 to -1.0] | -2.0 [-5.0 to -1.0]
  2nd to 5th MCP joints | -1.0 [-9.0 to 7.0] | 0.0 [-1.0 to 6.0] | -1.0 [-9.0 to 3.0]
  Total synovitis score | -3.0 [-9.0 to 9.0] | -1.0 [-5.0 to 3.0] | -3.0 [-10.0 to 0.0]

8. Secondary Outcome: Percent Change From Baseline to Week 12 in OMERACT RAMRIS Bone Erosion Score
Description: Bones from the wrist regions (carpal bones, distal radius, distal ulna and metacarpal bases) and the MCP joints (metacarpal heads and phalangeal bases) were assessed for erosion via MRI and scored separately based on the proportion of eroded bone compared to the 'assessed bone volume' judged from all available images. Scoring ranges from 0 (no erosion) to 10 (91-100%). For long bones, the 'assessed bone volume' is from the articular surface to a depth of 1 centimeter (cm) (if the articular surface is absent its best estimated position is used), and in carpal bones it is the whole bone. Results were summed, resulting in scores from 0 to 80 for the wrist region, 0 to 150 for the MCP joints, and 0 to 230 on aggregate. A negative value in change from Baseline score indicates an improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
percent change | -3.7 [-72.7 to 180.0] | 0.0 [-60.6 to 41.7]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided — Absolute Change in Bone erosion; Tocilizumab versus placebo. Since one-sided t-test was used all effects in the opposite direction of what was predicted have a p-value=1

9. Secondary Outcome: Absolute Change From Baseline to Week 12 in OMERACT RAMRIS Bone Erosion Score
Description: as for outcome 8
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
units on a scale | -0.5 [-16.0 to 10.0] | 0.0 [-20.0 to 5.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Test type: Superiority or Other; p = 1.00, t-test, 1 sided — Percentage Change in Bone erosion; Tocilizumab versus placebo. Since one-sided t-test was used all effects in the opposite direction of what was predicted have a p-value=1

10. Secondary Outcome: Percent Change From Baseline to Week 24 in OMERACT RAMRIS Bone Erosion Score
Description: Bones from the wrist regions (carpal bones, distal radius, distal ulna and metacarpal bases) and the MCP joints (metacarpal heads and phalangeal bases) were assessed for erosion via MRI and scored separately based on the proportion of eroded bone compared to the 'assessed bone volume' judged from all available images. Scoring ranges from 0 (no erosion) to 10 (91-100%). For long bones, the 'assessed bone volume' is from the articular surface to a depth of 1 cm (if the articular surface is absent its best estimated position is used), and in carpal bones it is the whole bone. Results were summed, resulting in scores from 0 to 80 for the wrist region, 0 to 150 for the MCP joints, and 0 to 230 on aggregate. A negative value in change from Baseline score indicates an improvement.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 7 | 9
percent change | -6.6 [-66.7 to 140.0] | -12.0 [-51.5 to 10.0] | -5.0 [-80.3 to 33.3]

11. Secondary Outcome: Absolute Change From Baseline to Week 24 in OMERACT RAMRIS Bone Erosion Score
Description: as for outcome 10
Time Frame: Week 24
Population: ITT population; participants from the placebo group who did not show an improvement of ≥ 20% in TJC and SJC were offered recovery therapy with tocilizumab 8mg/kg and were placed in Placebo-Tocilizumab 8mg/kg group.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 7 | 9
units on a scale | -1.5 [-9.0 to 7.0] | -2.0 [-17.0 to 1.0] | -2.0 [-15.0 to 4.0]

12. Secondary Outcome: Percent Change From Baseline to Week 12 in OMERACT RAMRIS Bone Edema Score
Description: Bones from the wrist regions (carpal bones, distal radius, distal ulna and metacarpal bases) and the MCP joints (metacarpal heads and phalangeal bases) were assessed for edema via MRI and scored separately based on the proportion of bone with edema. Scoring ranged from 0 to 3 as follows: 0: no edema; 1: 1-33% of bone edematous; 2: 34-66% of bone edematous; 3: 67-100%. Summing these values yielded a scale from 0-45 for the wrist region, 0-24 for the MCP joints, and 0-69 on aggregate.
Time Frame: Week 12
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
percent change | -17.1 [-100.0 to 66.7] | -15.0 [-83.3 to 137.5]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.266, t-test, 1 sided — Percentage Change in Bone oedema; Tocilizumab versus placebo

13. Secondary Outcome: Absolute Change From Baseline to Week 12 in OMERACT RAMRIS Bone Edema Score
Description: as for outcome 12
Time Frame: Week 12
Population: as for outcome 12
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
units on a scale | -3.0 [-19.0 to 7.0] | -2.0 [-25.0 to 11.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.337, t-test, 1 sided — Absolute Change in Bone edema; Tocilizumab versus placebo

14. Secondary Outcome: Percent Change From Baseline to Week 24 in OMERACT RAMRIS Bone Edema Score
Description: as for outcome 12
Time Frame: Week 24
Population: as for outcome 11
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 22 | 7 | 9
percent change | -37.5 [-100.0 to 6.7] | -37.5 [-100.0 to 10.7] | -51.9 [-85.2 to 116.7]

15. Secondary Outcome: Absolute Change From Baseline to Week 24 in OMERACT RAMRIS Bone Edema Score
Description: as for outcome 12
Time Frame: Week 24
Population: as for outcome 11
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 7 | 9
percent change | -5.5 [-29.0 to 1.0] | -3.0 [-9.0 to 3.0] | -10.0 [-23.0 to 7.0]

16. Secondary Outcome: Percent Change From Baseline to Week 12 in Dynamic Contrast Enhanced (DCE)-MRI Early Enhancement Rate (EER) Global Score
Description: Contrast enhancement was quantified in terms of initial rate of enhancement (IRE) and number of voxels (Nvox), which are extracted by examining individual signal intensity vs time curves derived from defined regions of interest (ROIs). A volume ROI was manually drawn around wrist and MCP 2-5 joints at each visit representative of size/volume of enhancement and underlying inflammation. Maximum enhancement (ME)=mean of ME and Nplateau+Nwashout (Nvoxels) are number of voxels that have a plateau and washout, used to assess volume of enhancing voxels within drawn ROIs. IRE=percentage increase of signal intensity (SI) until l ME is reached calculated as maximum increase in post-contrast SI divided by baseline SI; IRE=increase in SI in %/s from time of onset of enhancement to ME. EER reflects the IRE parameter and the output is the mean from all the assessed ROIs (range=between 0 and 1; 0=no change/enhancement, 1=maximum change/enhancement. Negative change from Baseline score=improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 12 | 9
percent change | -38.7 [-55.3 to -18.4] | -12.1 [-78.3 to 31.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.114, t-test, 1 sided — Percentage change in DCE-MRI EER (global); Placebo versus Tocilizumab

17. Secondary Outcome: Absolute Change From Baseline to Week 12 in Dynamic Contrast Enhanced (DCE)-MRI Early Enhancement Rate (EER) Global Score
Description: Contrast enhancement was quantified in terms of IRE and Nvox, which are extracted by examining individual signal intensity vs time curves derived from defined ROIs. A volume ROI was manually drawn around wrist and MCP 2-5 joints at each visit representative of size/volume of enhancement and underlying inflammation. ME=mean of ME and Nplateau+Nwashout (Nvoxels) are number of voxels that have a plateau and washout, used to assess volume of enhancing voxels within drawn ROIs. IRE=percentage increase of SI until l ME is reached calculated as maximum increase in post-contrast SI divided by baseline SI; IRE=increase in SI in %/s from time of onset of enhancement to ME. EER reflects the IRE parameter and the output is the mean from all the assessed ROIs (range=between 0 and 1; 0=no change/enhancement, 1=maximum change/enhancement. Negative change from Baseline score=improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 12 | 9
units on a scale | -0.002 [-0.004 to 0.001] | -0.001 [-0.01 to 0.002]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.239, t-test, 1 sided — Absolute Change in DCE-MRI EER; Tocilizumab versus placebo

18. Secondary Outcome: Percent Change From Baseline to Week 24 in DCE-MRI EER Global Score
Description: as for outcome 17
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 10 | 4 | 5
percent change | -45.4 [-68.6 to -11.8] | 23.0 [-37.5 to 76.5] | -32.7 [-57.6 to -3.5]

19. Secondary Outcome: Absolute Change From Baseline to Week 24 in DCE-MRI EER Global Score
Description: as for outcome 17
Time Frame: Week 24
Population: ITT population;
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 10 | 4 | 5
units on a scale | -0.003 [-0.01 to 0.00] | 0.0002 [0.00 to 0.01] | -0.002 [-0.01 to 0.00]

20. Secondary Outcome: Percent Change From Baseline to Week 12 in DCE-MRI EER MCP Score
Description: Contrast enhancement was quantified in terms of IRE and Nvox, which are extracted by examining individual signal intensity vs time curves derived from defined ROIs. A volume ROI was manually drawn around wrist and MCP 2-5 joints at each visit representative of size/volume of enhancement and underlying inflammation. ME=mean of ME and Nplateau+Nwashout (Nvoxels) are number of voxels that have a plateau and washout, used to assess volume of enhancing voxels within drawn ROIs. IRE=percentage increase of SI until l ME is reached calculated as maximum increase in post-contrast SI divided by baseline SI; IRE=increase in SI in %/s from time of onset of enhancement to ME. EER reflects the IRE parameter and the output is the mean from the MCP ROIs (range=between 0 and 1; 0=no change/enhancement, 1=maximum change/enhancement. Negative change from Baseline score=improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 10
percent change | -29.8 [-83.9 to 471.7] | -10.9 [-88.0 to 91.1]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.271, t-test, 1 sided — Percentage change in DCE-MRI EER (MCP); Placebo versus Tocilizumab

21. Secondary Outcome: Absolute Change From Baseline to Week 12 in DCE-MRI EER MCP Score
Description: as for outcome 20
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 10
units on a scale | -0.002 [-0.01 to 0.00] | -0.001 [-0.02 to 0.00]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.370, t-test, 1 sided — Absolute change in DCE-MRI EER (MCP); Placebo versus Tocilizumab

22. Secondary Outcome: Percent Change From Baseline to Week 24 in DCE-MRI EER MCP Score
Description: as for outcome 20
Time Frame: Week 24
Population: ITT population;
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 12 | 5 | 5
percent change | -32.3 [-100.0 to 40.0] | 15.0 [-56.9 to 45.7] | -29.1 [-66.8 to 7.5]

23. Secondary Outcome: Absolute Change From Baseline to Week 24 in DCE-MRI EER MCP Score
Description: as for outcome 20
Time Frame: Week 24
Population: ITT population;
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 12 | 5 | 5
units on a scale | -0.002 [-0.01 to 0.00] | 0.001 [0.00 to 0.01] | -0.001 [-0.01 to 0.00]

24. Secondary Outcome: Percent Change From Baseline to Week 12 in DCE-MRI EER Wrist Score
Description: Contrast enhancement was quantified in terms of IRE and Nvox, which are extracted by examining individual signal intensity vs time curves derived from defined ROIs. A volume ROI was manually drawn around wrist and MCP 2-5 joints at each visit representative of size/volume of enhancement and underlying inflammation. ME=mean of ME and Nplateau+Nwashout (Nvoxels) are number of voxels that have a plateau and washout, used to assess volume of enhancing voxels within drawn ROIs. IRE=percentage increase of SI until l ME is reached calculated as maximum increase in post-contrast SI divided by baseline SI; IRE=increase in SI in %/s from time of onset of enhancement to ME. EER reflects the IRE parameter and the output is the mean from the wrist ROIs (range=between 0 and 1; 0=no change/enhancement, 1=maximum change/enhancement. Negative change from Baseline score=improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 10
percent change | -24.8 [-81.6 to 102.1] | -19.1 [-84.3 to 111.4]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided — Percentage and absolute change in DCE-MRI EER (wrist); Placebo versus Tocilizumab

25. Secondary Outcome: Absolute Change From Baseline to Week 12 in DCE-MRI EER Wrist Score
Description: as for outcome 24
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 10
units on a scale | -0.002 [-0.01 to 0.00] | -0.001 [-0.01 to 0.00]

26. Secondary Outcome: Percent Change From Baseline to Week 24 in DCE-MRI EER Wrist Score
Description: as for outcome 24
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: percent change
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 12 | 5 | 5
percent change | -27.0 [-80.0 to 59.1] | 1.4 [-4.9 to 102.4] | -54.8 [-67.5 to -30.5]

27. Secondary Outcome: Absolute Change From Baseline to Week 24 in DCE-MRI EER Wrist Score
Description: as for outcome 24
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 12 | 5 | 5
units on a scale | -0.002 [-0.01 to 0.00] | 0.0001 [0.00 to 0.02] | -0.004 [-0.01 to 0.00]

28. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 was calculated from the number of swollen joints and tender joints (SJC and TJC) using the 28-joint count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and global health assessment (participant rated global assessment of disease activity using 10-mm visual analog scale [VAS]); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 12
Measure: Median (Full Range); unit: units on a scale
Groups:
- Placebo-Tocilizumab 8 mg/kg: Participants received placebo IV once every 4 weeks for a 12 weeks (total of 3 infusions). At 12 weeks, participants who did not respond to treatment (those who did not show improvement of ≥20% in TJC and SJC) received tocilizumab 8 mg/kg IV once every 4 weeks through Week 20.
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32 | 17 | 10
units on a scale
  Baseline (n=32,17,0) | 5.7 [3.4 to 8.0] | 6.2 [4.1 to 8.2] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks 16, 20, and 24.
  Week 12 (n=30,17,0) | 2.6 [1.1 to 5.8] | 5.6 [1.8 to 8.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks 16, 20, and 24.
  Week 24 (n=24,7,10) | 2.1 [0.8 to 4.1] | 3.9 [3.2 to 6.6] | 3.2 [1.5 to 5.1]

29. Secondary Outcome: Change From Baseline to Week 12 in DAS28 Global Score
Description: DAS28 was calculated from the number of swollen joints and tender joints (SJC and TJC) using the 28-joint count, the ESR (mm/hr) and global health assessment (participant rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. Change in DAS28 global score was determined as the difference in the scores at baseline and Week 12. A negative number indicated improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 15
units on a scale | -2.99 [-5.23 to -0.40] | 0.22 [-3.88 to 1.54]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

30. Secondary Outcome: Change From Baseline to Week 24 in DAS28 Global Score
Description: DAS28 was calculated from the number of swollen joints and tender joints (SJC and TJC) using the 28-joint count, the ESR (mm/hr) and global health assessment (participant rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. Change in DAS28 global score was determined as the difference in the scores at baseline and Week 24. A negative number indicated improvement.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 6 | 9
units on a scale | -3.4 [-6.5 to -1.8] | -1.2 [-5.0 to 0.6] | -2.9 [-4.1 to -1.5]

31. Secondary Outcome: Tender and Swollen Joint Counts
Description: TJC and SJC were determined using the 28 joint counts. Joints were classified as tender/not tender and swollen/not swollen and counted. The scores ranged from 0 to 28. Higher scores indicated higher disease activity.
Time Frame: Weeks 12 and 24
Population: as for outcome 12
Measure: Median (Full Range); unit: joints
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32 | 19 | 10
joints
  TJC, Week 12 (n=30,17,0) | 3.5 [0.0 to 28.0] | 8.0 [2.0 to 28.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks, 16, 20 and 24
  TJC, Week 24 (n=26,7,10) | 1.0 [0.0 to 7.0] | 7.0 [3.0 to 12.0] | 5.5 [0.0 to 12.0]
  SJC, Week 12 (n=30,17,0) | 1.5 [0.0 to 12.0] | 8.0 [0.0 to 24.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks, 16, 20 and 24
  SJC, Week 24 (n=26,7,10) | 0.0 [0.0 to 4.0] | 5.0 [1.0 to 17.0] | 2.5 [1.0 to 9.0]

32. Secondary Outcome: Change From Baseline to Week 12 in TJC
Description: Change in TJC was determined as the difference in the number of tender joints at baseline and the number at Week 12. A negative number indicated improvement.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: tender joints
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
tender joints | -6.5 [-17.0 to 0.0] | -2.0 [-16.0 to 10.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.067, t-test, 1 sided

33. Secondary Outcome: Change From Baseline to Week 24 in TJC
Description: Change in TJC was determined as the difference in the number of tender joints at baseline and the number at Week 24. A negative number indicated improvement.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: tender joints
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 26 | 7 | 10
tender joints | -8.5 [-26.0 to 0.0] | -5.0 [-21.0 to 0.0] | -7.5 [-22.0 to 0.0]

34. Secondary Outcome: Change From Baseline to Week 12 in SJC
Description: Change in SJC was determined as the difference in the number of swollen joints at baseline and the number at Week 12. A negative number indicated improvement.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: swollen joints
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
swollen joints | -7.0 [-19.0 to -1.0] | -1.0 [-13.0 to 10.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 1 sided

35. Secondary Outcome: Change From Baseline to Week 24 in SJC
Description: Change in SJC was determined as the difference in the number of swollen joints at baseline and the number at Week 24. A negative number indicated improvement.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: swollen joints
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 26 | 7 | 10
swollen joints | -8.5 [-23.0 to -2.0] | -7.0 [-21.0 to 1.0] | -5.0 [-8.0 to 0.0]

36. Secondary Outcome: Change From Baseline to Week 12 in Patient Global Assessment of Disease Activity
Description: General health was assessed using the Patient Global Assessment of Disease Activity, a 0 to 10 mm VAS, where 0 mm = very well and 10 mm = extremely bad. Participants were asked to answer the following question: "In general how would you rate your health over the last 2-3 weeks?". Participants responded by marking the line and the distance from the left edge was recorded.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: mm
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
mm | -3.8 [-9.4 to 2.0] | 0.2 [-6.6 to 6.8]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 1 sided

37. Secondary Outcome: Change From Baseline to Week 24 in Patient Global Assessment of Disease Activity
Description: as for outcome 36
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mm
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 26 | 7 | 10
mm | -4.4 [-9.5 to 2.6] | -1.5 [-7.1 to 3.7] | -1.4 [-5.4 to 1.0]

38. Secondary Outcome: Patient Global Assessment of Pain
Description: Patient's Global Assessment of Pain was assessed using a 10-mm horizontal VAS (0 to 10 mm) where 0=pain absent and 10=intolerable pain. Participants responded by placing a mark on the line to indicate their current level of pain; the distance from the left edge to the mark was recorded.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT population; n=number of participants assessed for the specific parameter at a given visit. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: mm
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32 | 19 | 10
mm
  Baseline (n=32,19,0) | 5.2 [2.6 to 10.0] | 5.1 [1.1 to 10.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks 16, 20, and 24.
  Week 4 (n= 31,18,0) | 3.2 [0.4 to 7.4] | 5.1 [1.3 to 10.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks 16, 20, and 24.
  Week 8 (n=31,17,0) | 2.8 [0.0 to 8.6] | 4.9 [1.9 to 8.3] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks 16, 20, and 24.
  Week 12 (n=30,17,0) | 2.2 [0.0 to 8.0] | 4.8 [1.0 to 8.6] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Weeks 16, 20, and 24.
  Week 16 (n=26,7,10) | 2.4 [0.0 to 6.6] | 3.8 [0.4 to 8.2] | 5.2 [1.5 to 8.8]
  Week 20 (n=26,7,10) | 1.5 [0.0 to 6.7] | 5.0 [2.0 to 6.5] | 3.8 [0.9 to 7.2]
  Week 24 (n=26,7,10) | 1.2 [0.0 to 8.0] | 5.3 [1.5 to 6.6] | 3.1 [0.7 to 6.2]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Test type: Superiority or Other; p < 0.001, Friedman's T test — Change from Baseline to Week 12
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.500, Friedman's T test — Change from Baseline to Week 12

39. Secondary Outcome: Change From Baseline to Week 12 in Patient Global Assessment of Pain
Description: Patient's Global Assessment of Pain was assessed using a 10-mm horizontal VAS (0 to 10 mm) where 0=pain absent and 10=intolerable pain. Participants responded by placing a mark on the line to indicate their current level of pain; the distance from the left edge to the mark was recorded. Change in Patient Global Assessment of Pain was determined as the difference in the scores at baseline and Week 12. A negative number indicated improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: mm
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 17
mm | -3.3 [-9.1 to 3.0] | -0.3 [-8.2 to 5.3]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.007, t-test, 1 sided

40. Secondary Outcome: Change From Baseline to Week 24 in Patient Global Assessment of Pain
Description: Patient's Global Assessment of Pain was assessed using a 10-mm horizontal VAS (0 to 10 mm) where 0=pain absent and 10=intolerable pain. Participants responded by placing a mark on the line to indicate their current level of pain; the distance from the left edge to the mark was recorded. Change in Patient Global Assessment of Pain was determined as the difference in the scores at baseline and Week 24. A negative number indicated improvement.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mm
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 26 | 7 | 10
mm | -3.7 [-9.4 to 2.8] | -3.4 [-4.4 to 3.2] | -1.5 [-5.9 to 1.9]

41. Secondary Outcome: Health Assessment Questionnaire - Disease Index (HAQ-DI) Scores
Description: The HAQ-DI includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0=without difficulties; 1=with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 12
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 32 | 19 | 10
units on a scale
  Global score, Baseline (n=30,16,0) | 2.1 [1.3 to 2.9] | 2.3 [1.4 to 2.9] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Global score, Week 12 (n=28,13,0) | 1.5 [1.0 to 2.5] | 2.3 [1.4 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Global score, Week 24 (n=26,7,10) | 1.3 [1.0 to 2.8] | 2.1 [1.6 to 2.5] | 2.1 [1.4 to 2.7]
  Dressing/grooming, Baseline (n=31,18,0) | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Dressing/grooming, Week 12 (n=30,16,0) | 1.0 [0.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Dressing/grooming, Week 24 (n=26,7,10) | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Arising, Baseline (n=32,19,0) | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Arising, Week 12 (n=30,17,0) | 1.0 [1.0 to 3.0] | 2.0 [0.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Arising, Week 24 (n=26,7,10) | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Eating, Baseline (n=26,14,0) | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Eating, Week 12 (n=27,10,0) | 2.0 [1.0 to 3.0] | 3.0 [2.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Eating, Week 24 (n=24,7,9) | 1.0 [1.0 to 3.0] | 3.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  Walking, Baseline (n=32,19,0) | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Walking, Week 12 (n=30,17,0) | 1.0 [0.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Walking, Week 24 (n=26,7,10) | 1.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0]
  Hygiene, Baseline (n=31,18,0) | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Hygiene, Week 12 (n=30,17,0) | 1.0 [0.0 to 3.0] | 2.0 [0.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Hygiene, Week 24 (n=26,7,10) | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Reach, Baseline (n=24,12,0) | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Reach, Week 12 (n=26,10,0) | 2.0 [0.0 to 3.0] | 2.0 [0.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Reach, Week 24 (n=23,7,8) | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 2.0] | 2.5 [1.0 to 3.0]
  Grip, Baseline (n=29,18,0) | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Grip, Week 12 (n=29,14,0) | 1.0 [0.0 to 3.0] | 2.0 [0.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Grip, Week 24 (n=26,7,9) | 1.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  Activity, Baseline (n=31,15,0) | 2.0 [1.0 to 3.0] | 2.0 [2.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Activity, Week 12 (n=29,14,0) | 2.0 [0.0 to 3.0] | 2.0 [0.0 to 3.0] | NA [NA to NA] — Data for the Placebo group with recovery therapy were collected only at Week 24.
  Activity, Week 24 (n=25,7,8) | 1.0 [1.0 to 3.0] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 3.0]

42. Secondary Outcome: Change From Baseline to Week 12 in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is an inflammatory marker and is used to assess disease activity in rheumatoid arthritis (RA). A reduction in ESR indicates improvement.
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: mm/hr
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 30 | 15
mm/hr | -19.0 [-93.0 to 0.0] | 2.0 [-49.0 to 39.0]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.001, t-test, 1 sided

43. Secondary Outcome: Change From Baseline to Week 24 in ESR
Description: ESR is an inflammatory marker and is used to assess disease activity in RA. A reduction in ESR indicates improvement.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mm/hr
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 6 | 9
mm/hr | -20.0 [-95.0 to 5.0] | -9.0 [-47.0 to 3.0] | -27.0 [-75.0 to -7.0]

44. Secondary Outcome: Change From Baseline to Week 12 in C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. CRP was measured in milligrams per deciliter (mg/dL).
Time Frame: Week 12
Population: ITT population. After Week 12, participants receiving placebo could have been switched to tocilizumab.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 29 | 15
mg/dL | -0.9 [-8.0 to 0.0] | -0.1 [-3.9 to 2.5]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 1 sided

45. Secondary Outcome: Change From Baseline to Week 24 in CRP
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 5 | 5
mg/dL | -1.2 [-8.0 to 0.0] | -0.2 [-2.9 to -0.02] | -0.6 [-9.7 to 0.0]

46. Secondary Outcome: Change From Baseline to Week 12 in Serum Cortisol
Description: Change in serum cortisol was determined as the difference in the scores at Baseline and Week 12.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 29 | 16
mg/dL | -1.4 [-53.0 to 102.3] | 2.5 [-31.6 to 119.3]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.118, t-test, 1 sided

47. Secondary Outcome: Change From Baseline to Week 24 in Serum Cortisol
Description: Change in serum cortisol was determined as the difference in the scores at Baseline and Week 24.
Time Frame: Week 24
Population: ITT population;
Measure: Median (Full Range); unit: mg/dL
Groups:
- Tocilizumab: Participants received tocilizumab 8 (minimum dose of 480 mg, maximum dose of 800 mg) IV once every 4 weeks for 24 weeks
- Placebo: Participants received placebo IV once every 4 weeks for a maximum of 24 weeks. At 12 weeks, participants who did not respond to treatment (those who did not show improvement of at least 20% in tender joint count and swollen joint count) were offered rescue therapy with open-label tocilizumab 8 mg/kg every 4 weeks.
- Placebo-Tocilizumab: At 12 Weeks participants who did not show an improvement of ≥20% in tender and swollen joint counts were offered a rescue therapy with open-label tocilizumab 8mg/kg every 4 weeks
Arm/Group | Tocilizumab | Placebo | Placebo-Tocilizumab
Number analyzed (Participants) | 25 | 7 | 10
mg/dL | -2.5 [-40.1 to 51.8] | -5.2 [-32.0 to 6.0] | -5.1 [-63.2 to 106.2]

48. Secondary Outcome: Change From Baseline to Week 12 in Plasma Adrenocorticotrophic Hormone (ACTH)
Description: Change in Plasma ACTH was determined as the difference in the scores at Baseline and Week 12.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 28 | 15
mg/dL | 0.00 [-10.27 to 7.41] | 0.00 [-7.62 to 4.67]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided

49. Secondary Outcome: Change From Baseline to Week 24 in Plasma ACTH
Description: Change in plasma ACTH was determined as the difference in the scores at baseline and Week 24.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Groups:
- Placebo-Tocilizumab 8 mg/kg: Patient's Global Assessment of Pain was assessed using a 10-mm horizontal VAS (0 to 10 mm) where 0=pain absent and 10=intolerable pain. Participants responded by placing a mark on the line to indicate their current level of pain; the distance from the left edge to the mark was recorded. Change in Patient Global Assessment of Pain was determined as the difference in the scores at baseline and Week 12. A negative number indicated improvement.
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 6 | 10
mg/dL | -0.4 [-13.7 to 12.7] | -0.3 [-2.0 to 0.0] | 0.8 [-1.9 to 4.1]

50. Secondary Outcome: Change From Baseline to Week 12 in Serum Androstenedione
Description: Change in serum androstenedione was determined as the difference in the scores at Baseline and Week 12.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 28 | 16
mg/dL | 0.01 [-0.57 to 0.29] | 0.01 [-0.12 to 0.18]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.437, t-test, 1 sided

51. Secondary Outcome: Change From Baseline to Week 12 in 17 Hydroxy Progesterone (17OHP)
Description: Change in 17OHP was determined as the difference in the scores at Baseline and Week 12.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 28 | 15
mg/dL | -0.01 [-1.90 to 1.86] | -0.03 [-0.60 to 0.12]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 1.00, t-test, 1 sided

52. Secondary Outcome: Change From Baseline to Week 24 in Serum Androstenedione
Description: Change in serum androstenedione was determined as the difference in the scores at Baseline and Week 24.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 25 | 6 | 10
mg/dL | 0.02 [-1.56 to 0.70] | 0.01 [-0.10 to 0.06] | -0.002 [-0.71 to 0.36]

53. Secondary Outcome: Change From Baseline to Week 24 in 17OHP
Description: Change in 17OHP was determined as the difference in the scores at Baseline and Week 24.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 23 | 6 | 10
mg/dL | -0.01 [-1.97 to 1.03] | -0.07 [-0.86 to 0.46] | -0.02 [-0.50 to 0.20]

54. Secondary Outcome: Change From Baseline to Week 12 in Serum Dehydroepiandrosterone (DHEA)
Description: Change in DHEA was determined as the difference in the scores at Baseline and Week 12.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 28 | 15
mg/dL | -0.07 [-6.09 to 2.90] | 0.00 [-5.87 to 4.03]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.190, t-test, 1 sided

55. Secondary Outcome: Change From Baseline to Week 24 in Serum DHEA
Description: Change in DHEA was determined as the difference in the scores at Baseline and Week 24.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 6 | 10
mg/dL | 0.17 [-5.67 to 4.07] | -0.73 [-3.45 to 2.50] | 0.40 [-10.43 to 3.38]

56. Secondary Outcome: Change From Baseline to Week 12 in Neuropeptide Y
Description: Change in Neuropeptide Y was determined as the difference in the scores at Baseline and Week 12.
Time Frame: Week 12
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo
Number analyzed (Participants) | 29 | 16
mg/dL | -13.3 [-91.4 to 60.3] | -0.7 [-45.4 to 51.2]
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.051, t-test, 1 sided

57. Secondary Outcome: Change From Baseline to Week 24 in Neuropeptide Y
Description: Change in Neuropeptide Y was determined as the difference in the scores at Baseline and Week 24.
Time Frame: Week 24
Population: ITT population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Number analyzed (Participants) | 24 | 6 | 9
mg/dL | -11.1 [-80.8 to 80.6] | -2.5 [-44.5 to 58.4] | -13.9 [-52.8 to 28.2]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the day of screening until the end of study at Week 24.
Arm/Group | Tocilizumab 8 mg/kg | Placebo | Placebo-Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/35 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 29/35 | 7/10 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=35) | Placebo (N=10) | Placebo-Tocilizumab 8 mg/kg (N=9)
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gluteal cleft cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=35) | Placebo (N=10) | Placebo-Tocilizumab 8 mg/kg (N=9)
Hepatotoxicity (Hepatobiliary disorders) | 2 | 2 | 0
Hypercholesterolemia (Investigations) | 3 | 1 | 1
Urinary Tract infection (Infections and infestations) | 4 | 1 | 0
Malar rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Hepatic toxicity (Hepatobiliary disorders) | 2 | 2 | 0
Abnormal liver function tests (Investigations) | 0 | 1 | 0
Liver Enzyme Elevation (Investigations) | 2 | 0 | 0
Elevated ALT (Investigations) | 2 | 0 | 0
Transaminase Elevation (Investigations) | 1 | 0 | 0
Bilirubin Elevation (Investigations) | 1 | 0 | 0
Back pain (General disorders) | 1 | 0 | 0
Blood Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Cough (General disorders) | 1 | 0 | 1
Dislipidemia (Investigations) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Epigastric pain (Gastrointestinal disorders) | 1 | 0 | 0
Facial paralysis on the right side (Nervous system disorders) | 1 | 0 | 0
Fall (General disorders) | 1 | 0 | 0
Finger cut (General disorders) | 1 | 0 | 0
Flu (Infections and infestations) | 2 | 0 | 0
Hematoma cyclid of the right eye (Blood and lymphatic system disorders) | 1 | 0 | 0
Herpes simplex in the lips (Infections and infestations) | 1 | 0 | 0
Hoarseness (General disorders) | 1 | 0 | 0
Hypertriglyceridemia (Investigations) | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0
Infected traumatic right leg ulcer (Infections and infestations) | 1 | 0 | 0
Inter-digital wound (General disorders) | 1 | 0 | 0
Left leg cellulitis (General disorders) | 1 | 1 | 0
Leg ulcer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mild renal failure (Renal and urinary disorders) | 1 | 0 | 0
Nausea (General disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Oral aftosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Tooth ache (General disorders) | 1 | 0 | 0
Upper airways infection (Infections and infestations) | 1 | 0 | 0
Vaginal labial folliculitis (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Flu-like syndrome (General disorders) | 0 | 1 | 1
Nitritis Elevation (Investigations) | 0 | 1 | 0
Odynophagia (General disorders) | 0 | 1 | 0
Urine Leukocyte elevation (Blood and lymphatic system disorders) | 0 | 1 | 0
Varicose vein rupture (Blood and lymphatic system disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gingivorrhagea in patient with low platelets (General disorders) | 0 | 0 | 1
Mouth mucositis (Infections and infestations) | 0 | 0 | 1
Sputum (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.